CLINICAL TRIAL: NCT03574636
Title: Optical Coherence Tomography Compared With Intravascular Ultrasound or Quantitative Coronary Analysis to Guide Stent Implantation in the Treatment of Moderate-to-severe Calcified Lesion in Coronary Artery
Brief Title: OCT vs IVUS vs QCA to Guide Moderate-to-severe Calcified Lesion Stent Implantation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai MicroPort Medical (Group) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TARGET 3C
Record Dates: First submitted 2018-06-20; First posted 2018-07-02 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Optical Coherence Tomography; Intravascular Ultrasound; Angiography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- OCT guidance (Active Comparator): Firehawk stent implantation will be performed with Optical Coherence Tomography guidance.
  At the end of the procedure, a final DSA imaging run and OCT measurement must be performed.
  At 13-month follow-up, DSA imaging run must be performed. At 3-month follow-up, OCT imaging run must be performed in the first 66 consecutive patients.
  Interventions: Device: OCT guidance
- IVUS guidance (Active Comparator): Firehawk stent implantation will be performed with Intravascular Ultrasound guidance.
  At the end of the procedure, a final DSA imaging run and OCT measurement must be performed.
  At 13-month follow-up, DSA imaging run must be performed. At 3-month follow-up, OCT imaging run must be performed in the first 66 consecutive patients.
  Interventions: Device: IVUS guidance
- QCA guidance (Active Comparator): Firehawk stent implantation will be performed with Intravascular Ultrasound guidance.
  At the end of the procedure, a final DSA imaging run and OCT measurement must be performed.
  At 13-month follow-up, DSA imaging run must be performed. At 3-month follow-up, OCT imaging run must be performed in the first 66 consecutive patients.
  Interventions: Device: QCA

INTERVENTIONS:
Device: OCT guidance — OCT guide stent implantation
  Arms: OCT guidance
Device: IVUS guidance — IVUS guide stent implantation
  Arms: IVUS guidance
Device: QCA — QCA guide stent implantation
  Arms: QCA guidance

SUMMARY:
This study is a prospective, multi-center, randomized controlled clinical trial, aims to assess the safety and effectiveness of Optical Coherence Tomography or Intravascular Ultrasound or Quantitative Coronary Analysis to guide Firehawk stent implantation , and compared the treatment of moderate-to-severe calcified lesion in coronary artery.

DETAILED DESCRIPTION:
This clinical trial will enroll 375 subjects and assign to groups in a 1:1:1 ratio (base on Intravascular Ultrasound [IVUS]-guided treatment group : Optical Coherence Tomography [OCT]-guided treatment group : Quantitative Coronary Angiography [QCA]-guided treatment group) who have moderate-severe calcified lesions in de novo native coronary artery with ≥2.50 mm to ≤4.00 mm in diameter (visual measurement) from a maximum of 25 study sites in China. After the stent is implanted satisfactorily, OCT examinations will be performed on the subjects of these three groups to observe stent expansion after implantation. At 13 months after procedure, all subjects will receive QCA examination.

OCT sub-group study: The initial 66 ongoing subjects from the three treatment groups (IVUS-guided treatment group : OCT-guided treatment group : QCA-guided treatment group) who provided informed consent and successfully randomized will receive OCT examinations at three months follow up after baseline procedure.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be 18 to 80 years age
* Subject (or legal guardian) understands the trial requirements and the treatment procedures and provides written informed consent before any trial-specific tests or procedures are performed;
* Subject is eligible for percutaneous coronary intervention (PCI);
* Subject has symptomatic coronary artery disease with objective evidence of ischemia or silent ischemia (including NST-ACS, stable CAD and STEMI（duration over 4 weeks）);
* Subjects are eligible candidates for coronary artery bypass graft surgery (CABG);
* Left ventricular ejection fraction (LVEF) detected by cardiac ultrasound within 30 days ≥ 30%;
* Subject is willing to comply with all protocol-required follow-up evaluation.

Angiographic Inclusion Criteria (visual estimate):

* The target lesion must be a new lesion and has moderate-to-severe calcification which located in a visually estimated reference diameter ≥2.5 mm and ≤4.0 mm in native coronary artery;
* Target lesion diameter stenosis ≥70% and ≤99%
* Target lesion length ≤70mm
* Judgment of moderate-to-severe calcification:

  * Grade II (moderate) calcification:

Before angiography with or without contrast agent injected, the opacity and deformation of coronary artery can be basically seen, the contour of coronary artery can be basically seen and the contrast agent can fully cover the opacity of blood vessel

* Grade III (severe) calcification:

Before angiography with or without contrast agent injected, the opacity and deformation of coronary artery can be basically seen, the contour of coronary artery is clearly visible and the contrast agent can partially cover the opacity of blood vessel

* Grade IV (extremely severe) calcification:

Before angiography with or without contrast agent injected, the opacity of coronary artery can be clearly seen, the contour and deformation are completely visible, and whether the contrast agent is injected is not highly correlated with the changes in the opacity density of blood vessel.

Exclusion Criteria:

* Subjects recently suffer from STEMI (within 4 week), and ECG changes/clinical symptoms consistent with AMI or accompanied with increased cardiac biomarkers (CK-MB, CK, TNT or TNI) , and if any of the following criteria is meet in the procedure, patients are excluded; CK-MB> 2ULN, regardless of the value of total CK; total CK> 2ULN, CK-MB or Tn is abnormal;

If CK-MB or CK was not detected, but cTN> 1ULN, and at least one of the following:

schemic symptoms and ECG changes of new ischemia; Development of pathologic Q waves in the ECG; Imaging evidence of new loss of viable myocardium or new regional wall motion abnormality.

* Subject with hemodynamic instability or severely decreased activity tolerance (KILLIP classification >2 or NYHA classification >2 );
* Severely ejection fraction reduced heart failure ( LVEF < 30%)
* Subjects were detected ventricular aneurysm greater than 3.0*2.0cm or intraventricular thrombosis by cardiac ultrasonography in 30 days;
* Subjects had an organ transplant or are waiting for an organ transplant;
* Subjects are receiving chemotherapy or will receive a chemotherapy within 30 days after PCI;
* Subjects are undergoing chronic (over 72 hours) anticoagulant therapy (such as heparin and coumarin) other than acute coronary syndrome;
* Subjects have confirmed or suspected liver disease, including hepatitis lab results;
* Subjects with elevated serum creatinine level >3.0mg/dL or undergoing dialysis therapy
* Subjects with active peptic ulcer, active gastrointestinal (GI) bleeding or other bleeding diathesis or coagulopathy, or refused a blood transfusion;
* Subjects with cerebral vascular accident (CVA) or transient ischemic attack (TIA) in the past 6 months, or with permanent nerve defects;
* Subjects had any PCI (such as balloon angioplasty, stent, cutting balloon,atherectomy) treatment in target vessels (including collateral) within 13 months prior to baseline;
* Within10mm proximal or distal to the target lesion (including branch artery) had received any PCI prior to baseline;
* Non target vessel had got any PCI in 24 hours prior to baseline;
* Subjects plan to undergo PCI or CABG in 13 months after the baseline PCI;
* Subjects have any coronary endovascular brachytherapy treatment previously;
* Subjects associated with drugs allergy (such as sirolimus, or structure-related compounds fluorinated polymers, thiophenepyridine or aspirin);
* Subjects are suffering from other serious illness (such as cancer, congestive heart failure), which may cause drop in life expectancy to less than 13 months;
* Subjects are currently abusing drugs (such as alcohol, cocaine, heroin, etc);
* Subject plan to undergo any operations that may lead to confuse with the programme;
* Subjects were participating in another study of drug or medical device which did not meet its primary endpoint;
* Subjects plan to pregnant within 13 months after baseline;
* Subjects are pregnant or breastfeeding women.

Angiographic Exclusion Criteria (visual estimate):

* Target lesions with the following criteria:

More than 2 target vessel and 2 target lesion Left main Ostial lesion Bifucation lesion( stenosis >70%), branch vessel diameter ≥2.5 mm and lesion length more than 5mm Target lesion located in saphenous vein grafts or arterial grafts Via saphenous vein grafts or arterial graft to treat the target lesion Thrombosis in target lesion Endomembrane tear in target lesion Restenosis in stent prior to the procedure Chronic total occlusion

* Subjects with unprotected left main coronary artery disease (diameter stenosis >50%);
* Subjects have a protected left main coronary artery disease (diameter stenosis> 50% and left coronary artery bypass surgery), as well as target lesions located in the LAD and LCX;
* Subjects with other lesions of clinical significance, may be need intervention within 13 months after baseline.
* Either reason (ig. severe tortuosity, etc) causing stent improperly placed and positioned

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 375 (Estimated)
Dates: Start 2019-10-18 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
in-stent late loss | 13 months
  the difference between the minimal lumen diameter immediately after stent implantation and the minimal lumen diameter by angiography review 13 months after the procedure

SECONDARY OUTCOMES:
instant Minimum Stent Area (MSA) | during PCI procedure
  instant Minimum Stent Area (MSA) measured by Optical Coherence Tomography (OCT) during PCI procedure
stent neointimal thickness | 3 months
  stent neointimal thickness at 3 months measured by Optical Coherence Tomography (OCT)

OTHER OUTCOMES:
Target Vessel Revascularization (TVR) | In hospital and at 30 days, 3, 6, 12 ,13 months and 2-5 years after index procedure
Target Vessel Failure (TVF) | In hospital and at 30 days, 3, 6, 12 ,13 months and 2-5 years after index procedure
  Combined endpoints of Cardiac death, myocardial infarction (MI) and ischemia-driven Target Vessel Revascularization (TVR)
Target Lesion Revascularization (TLR) | In hospital and at 30 days, 3, 6, 12 ,13 months and 2-5 years after index procedure
  Defined as any repeat percutaneous coronary intervention (PCI) of the target lesion or bypass surgery for restenosis or other complication of the target lesion.
Target Lesion Failure (TLF) | In hospital and at 30 days, 3, 6, 12 ,13 months and 2-5 years after index procedure
  Combined endpoints of Cardiac death, myocardial infarction (MI) and ischemia-driven Target Lesion Revascularization (TLR)

CONTACTS AND LOCATIONS:
Overall Officials: Yundai Chen, MD, Principal Investigator — The General Hospital of People's Liberation Army(301 hospital)
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China